CLINICAL TRIAL: NCT05845385
Title: Comparison of Lumbar Epidural Analgesia, Transversus Abdominis Plane Block and Wound Infiltration for Postoperative Pain Relief in Major Abdominal Gynecological Surgery
Brief Title: Postoperative Pain Relief After Major Abdominal Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Hakki Unlugenc, professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAS
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Pain
Keywords: epidural analgesia; pain score; morphine; transversus abdominis plane block; wound infiltration
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lumbar epidural analgesia with bupivacaine (Active Comparator): For postoperative analgesia; Lumbar epidural catheter inserted at L3-4 or L4-5 epidural space before anesthesia induction in the sitting position. After the end of surgery but approximately 20 minutes before extubation, 0.125% bupivacaine 20 ml administered through epidural catheter and the catheter was removed.
  Interventions: Procedure: lumbar epidural analgesia with bupivacaine
- transversus abdominis plane block with bupivacaine (Active Comparator): For postoperative analgesia; After the end of surgery but before extubation, USD-guided TAP block was performed with 0.125% bupivacaine 20 ml to the anatomic neurofacial space between the internal oblique and transersus abdominis muscles, bilaterally (10 ml for each side).
  Interventions: Procedure: transversus abdominis plane block with bupivacaine
- wound infiltration with bupivacaine (Active Comparator): For postoperative analgesia; After the end of surgery but before extubation, 0.125% bupivacaine 20 ml administered to the surgical incision site.
  Interventions: Procedure: wound infiltration with bupivacaine

INTERVENTIONS:
Procedure: lumbar epidural analgesia with bupivacaine — postoperative analgesic method
  Arms: lumbar epidural analgesia with bupivacaine
Procedure: transversus abdominis plane block with bupivacaine — postoperative analgesic method
  Arms: transversus abdominis plane block with bupivacaine
Procedure: wound infiltration with bupivacaine — postoperative analgesic method
  Arms: wound infiltration with bupivacaine

SUMMARY:
The aim of our study was to compare the effects of Lomber Epidural Analgesia (LEA), Transversus Abdominis Plane (TAP) block and Local Anesthetic Infiltration (LAI) on postoperative morphine consumption, time to first recue analgesic request, pain and patient satisfaction scores and side effects were compared in the patients undergoing major gynecologic/oncology lower abdominal surgery.

DETAILED DESCRIPTION:
Following faculty ethical committee approval and written informed consent, 81 patients were included in our prospective, randomized and double-blind study. Patients were divided into 3 groups: lumbar epidural block (Group E), TAP block (Group T), and wound infiltration (Group I). Demographic data, surgical characteristics, hemodynamic values, pain scores at rest and on movement, morphine consumption, additional analgesic requirement, side effects at 1, 2, 6, 12, 24, 36 and 48th hours after surgery, and patient satisfaction scores at 24 and 48th hours were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II,
* between the age of 18-69,
* undergoing major gynecological abdominal surgery under general anesthesia

Exclusion Criteria:

* lack of patient consent
* ASA > III
* sensitivity or contraindication to study drugs
* conditions in which epidural anesthesia is contraindicated
* emergency and urgent surgery
* inability to comprehend pain scale
* any contraindication to the use of patient controlled analgesia (PCA) device.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study was conducted on female patients undergoing major abdominal gynecological surgery.
Enrollment: 81 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
morphine consumption | change from baseline morphine comsumption at 48 hours
  At the end of the surgery, the patients were allowed to use the patient controlled analgesia device (PCA). The PCA (CADD Legacy PCA pump, Smiths Medical MD, Inc. St. Paul, MN) was prepared with 40 mg morphine HCl in 100 ml saline. The PCA doses of morphine consisted of a bolus dose of 0.02 mg/kg every 15 minutes without a background infusion. Morphine consumption (mg) was evaluated and recorded postoperative 48 hours.

SECONDARY OUTCOMES:
pain scores | change from baseline pain scores at 48 hours
  postoperative pain scores of the patients were recorded using visual analog scale (VAS; 0=no pain, 10=worst pain)
patient satisfaction score | postoperative 24 and 48 hours
  patient satisfaction scores were recorded using patient satisfaction scale (0= worst, 10=excellent)
time to first rescue analgesic | postoperative 48 hours
  If the patients complained of pain despite the analgesia regimen, iv 50 mg meperidine was given as a rescue analgesic.
side effects | postoperative 48 hours
  all patients were visited after surgery in the ward and side effects were evaluated and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Hakkı - Unlugenc, Proffessor, Study Chair — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)